CLINICAL TRIAL: NCT06033651
Title: Long Term Follow up of the Titanium Modular Revision Hip System up (TinT 10)
Brief Title: Long Term Follow up of the Titanium Modular Revision Hip System up (TinT 10) Levels
Acronym: TinT10
Status: Not yet recruiting | Type: Observational
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: RL1 879
Record Dates: First submitted 2023-08-29; First posted 2023-09-13 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Hip Surgery
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Only 1 arm for the study: All participants shall receive the same treatment.
  Interventions: Radiation: x-ray

INTERVENTIONS:
Radiation: x-ray — AP view of pelvis
  Other Names: AP view of pelvis

SUMMARY:
Patients are to be approached to attend clinic who have been identified as being implanted with either a Lima Corporate Delta Revision TT, Delta One TT or the Delta Multihole Systems hip systems between 2011 and 2015, a minimum of 10 years since hip surgery. They will be x-rayed (AP pelvis and a lateral view) and have a clinical review in clinic.

DETAILED DESCRIPTION:
Since its popularisation in the 1960's, Hip replacements have become one of the NHS's highest volume procedures. Unfortunately, hip replacements can fail with on average 8,500 revision hip replacements being performed each year pre-covid(1). Often this is very complex with destruction of the normal anatomy leaving surgeons with a significant challenge in ensuring appropriate positioning of the socket within the confines of the patient's anatomy.

The Lima Corporate Delta systems are designed to help surgeons with this very problem by providing the option of a 'face changer' allowing surgeons to place a socket within a socket.

To allow for this function, the 'face changer' must connect with the acetabular cup (socket).

140 patients have been identified as having had this modular acetabular system implanted at the RJAH in 2012 & 2014, going into 2015. The aim of this study is to therefore identify the survivorship of these implants at 10 years.

ELIGIBILITY:
Inclusion Criteria:

All adult patients who had Lima Corporate modular titanium acetabular component implants implanted between 2011 and 2015.

Exclusion Criteria:

Deceased patients Patients who have undergone a subsequent acetabular revision Patients that lack capacity Prisoners in the custody of HM Prison service or who are offenders supervised by the probation service in England or Wales.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients who had Lima Corporate modular titanium acetabular component implants implanted between 2011 and 2015.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-10 (Estimated); Primary Completion 2026-05-14 (Estimated); Study Completion 2026-05-14 (Estimated)

PRIMARY OUTCOMES:
The survivourship of the modular acetabular hip system at 10 years post-op | Participants will be invited to attend a one time clinic visit, after which their participation in the study has ended.
  This study will be the largest study to look at the survivorship of this acetabular system. Survivorship will be to the point of revision and clinical outcome survivorship is to the point of radiological loosening and PROMs data collection.

CONTACTS AND LOCATIONS:
Overall Officials: Robin Banerjee, Principal Investigator — The Robert Jones and Agnes Hunt Orthopaedic Hospital Foundation Trust

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ben-Shlomo Y, Blom A, Boulton C, Brittain R, Clark E, Dawson-Bowling S, Deere K, Esler C, Espinoza O, Evans J, Goldberg A, Gregson C, Howard P, Jameson S, Jennison T, Judge A, Lawrence S, Lenguerrand E, Marques E, McCormack V, Newell C, Pegg D, Penfold C, Porter M, Price A, Reed M, Rees J, Royall M, Sayers A, Stonadge J, Swanson M, Taylor D, Toms A, Watts A, Whitehouse M, Wilkinson M, Wilton T, Young E. The National Joint Registry 19th Annual Report 2022 [Internet]. London: National Joint Registry; 2022 Oct. Available from http://www.ncbi.nlm.nih.gov/books/NBK587525/ PMID 36516281
- [Background] Liu TK, Liu SH, Chang CH, Yang RS. Concentration of metal elements in the blood and urine in the patients with cementless total knee arthroplasty. Tohoku J Exp Med. 1998 Aug;185(4):253-62. doi: 10.1620/tjem.185.253. PMID 9865472